CLINICAL TRIAL: NCT00839176
Title: A Double-blinded, Randomized, Placebo-controlled, Dose-Exploring Study of RX-10100 When Given for Eight Consecutive Weeks to Subjects With Major Depression Disorder (MDD)
Brief Title: Efficacy Study of RX-10100 to Treat Major Depressive Disorder (MDD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rexahn Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RX-10100-P2A-002
Record Dates: First submitted 2009-02-05; First posted 2009-02-09 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-11

CONDITIONS: Major Depressive Disorder (MDD)
Keywords: Major Depressive Disorder (MDD); Serdaxin; Rexahn
MeSH Terms: conditions — Depressive Disorder, Major | interventions — RX-10100

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Placebo (w/o API)
  Interventions: Drug: RX-10100
- 2 (Experimental): 5mg dose of RX-10100
  Interventions: Drug: RX-10100
- 3 (Experimental): 10mg dose of RX-10100
  Interventions: Drug: RX-10100
- 4 (Experimental): 15 mg dose of RX-10100
  Interventions: Drug: RX-10100

INTERVENTIONS:
Drug: RX-10100 — Extended-release tablet, 5~15mg, twice day (morning & evening) at least 30 min before meal, 8 weeks
  Other Names: Serdaxin

SUMMARY:
The primary objective of this Phase IIa trial is to determine the effective dose and treatment period for an upcoming RX-10100 Phase IIb trial in subjects with major depression disorder (MDD). The secondary objectives of this trial are to evaluate the safety and quality of life in subjects with MDD receiving RX-10100 treatment.

ELIGIBILITY:
Inclusion Criteria:

* Males or females between 18 and 65 years old
* Diagnosis of MDD using DSM-IV criteria
* Have a score of 20 or more on the HAM-D-17
* Have a score of 4 or more on the CGI-S
* Written informed consent obtained
* Have a negative serum (P-HCG) pregnancy test at screening (for all women)
* Female subjects must meet one of the following criteria: (a) Be surgically sterile or (b) Agree that, if sexually active they will use oral contraceptives, double barrier contraception (E.g., condom with spermicide), intrauterine device, or other method approved by the sponsor.

Exclusion Criteria:

* Have a BMI > 40 or < 18
* Unstable angina pectoris
* History of myocardial infarction, stroke, or life-threatening arrhythmia within the prior 6 months
* Uncontrolled atrial fibrillation/flutter at screening
* Severe chronic or acute liver disease; history of moderate or severe hepatic impairment
* Clinically significant chronic hematological disease which may lead to priapism, such as sickle cell anemia and leukemia
* Bleeding disorder
* Resting hypotension or hypertension
* History of malignancy (cancers) within the past 5 years (other than squamous or basal cell skin cancer)
* NYHA Class III or IV heart failure
* Substance abuse/dependence within the past 6 months
* Significant suicidal ideation based on the C-SSRS
* Other current nondepressive Axis I disorders
* Depressive episode duration of less than 1 month or greater than 9 months
* Bipolar disorder
* Dysthmic disorder
* Borderline personality disorder
* Psychotic disorder/current psychotic features
* Any abnormal findings on the screening ECG judged clinically significant by the Investigator
* Any medical condition that is not stabilized or is anticipated to require hospitalization within 6 months, in the opinion of the Investigator
* Any history of cholestatic jaundice or liver cirrhosis
* Hyper- or hypothyroidism unless the subject has received a stable dose of thyroid medication for at least 3 months prior to the screening visit
* Women, who are breast-feeding, have been lactating within 3 months prior to screening
* Concurrent psychotherapy
* Subjects who have received any other investigational drug (including placebo) within 30 days before Visit 1
* Use of any treatment for MDD within 7 days of Visit 1 (14 days for fluoxetine) and during the study other than the study medication
* Use of antidepressants, anxiolytics, or other psychoactive drugs within 14 days of Visit 1 and during the study
* Concomitant use of antibiotics in the penicillin class (for the reduction of the potential for any additive or synergistic hepatotoxicity)
* A positive urine drug screen
* Elevation of AST and/or ALT > 3 times the upper limit of normal (ULN)
* Diabetic subjects with an HbAlc ≥ 12%
* Any abnormal screening laboratory values judged clinically significant by the Investigator
* Previous nonresponse or hypersensitivity to two or more trials of antidepressant medication given in adequate doses and duration for the treatment of symptoms present in the current illness
* Subjects with known hypersensitivity to any antibiotic in the penicillin class
* Subjects who are illiterate or unable to understand the questionnaires
* Subjects who, in the opinion of the investigator, would be non-compliant with the visit schedule of study procedures
* Subjects who pose potential harm to others

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2009-01; Primary Completion 2009-09 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline at 8 weeks on the Montgomery-Asberg Depression Rating Scale (MADRS) | 8 weeks

SECONDARY OUTCOMES:
Changes from baseline on the HAM-D | 8 weeks
Changes from baseline on the QIDS-SR | 8 weeks
CGI-I scale at the end of treatment, | 8 weeks
Side effects during and immediately following the treatment period | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Christine Peterson, PhD, Study Director — Rexahn Pharmaceuticals, Inc.
Locations (3):
- United States (3):
  - Denver, Colorado
  - Atlanta, Georgia
  - Rockville, Maryland

REFERENCES:
- [Derived] Riesenberg R, Rosenthal J, Moldauer L, Peterson C. Results of a proof-of-concept, dose-finding, double-blind, placebo-controlled study of RX-10100 (Serdaxin(R)) in subjects with major depressive disorder. Psychopharmacology (Berl). 2012 Jun;221(4):601-10. doi: 10.1007/s00213-011-2604-x. Epub 2011 Dec 28. PMID 22203317